CLINICAL TRIAL: NCT00096304
Title: Phase I Trial of Epirubicin and Taxotere in Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Epirubicin and Docetaxel in Treating Patients With Metastatic Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MUSC-100781; CDR0000378045 (Registry Identifier: PDQ (Physician Data Query)); MUSC-HR-11325; AVENTIS-MUSC-100781
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: docetaxel
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of epirubicin when given with docetaxel in treating patients with metastatic prostate cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Meets 1 of the following criteria:

  * Measurable disease with any prostate-specific antigen (PSA) value

    * Unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
    * Histologic confirmation required if measurable disease is confined to a solitary lesion
  * Non-measurable disease with PSA ≥ 5 ng/mL*

    * The following are considered non-measurable disease:

      * Bone lesions
      * Pleural or pericardial effusion
      * Ascites
      * CNS lesions
      * Leptomeningeal disease
      * Irradiated lesions unless disease progression was documented after prior radiotherapy NOTE: *Patients with PSA ≥ 5 ng/mL only are not eligible
* Progressive systemic disease despite ≥ 1 prior standard endocrine therapy with orchiectomy, luteinizing hormone-releasing hormone (LHRH) agonist, or diethylstilbestrol, as indicated by 1 of the following criteria:

  * Objective evidence of increase > 20% in the sum of the longest diameters of target lesions from the time of maximal regression OR the appearance of 1 or more new lesions
  * One or more new lesions on bone scan secondary to prostate cancer AND PSA ≥ 5 ng/mL
  * Elevated PSA (≥ 5 ng/mL) with 2 consecutive increases from baseline (taken ≥ 1 week apart)
* Serum testosterone ≤ 50 ng/dL for patients without bilateral orchiectomy

  * Patients who have not had a bilateral orchiectomy should continue therapy with primary testicular androgen suppression (e.g., LHRH analogues)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Meets 1 of the following criteria:

  * AST or ALT normal AND alkaline phosphatase ≤ 5 times upper limit of normal (ULN)
  * AST or ALT ≤ 1.5 times ULN AND alkaline phosphatase ≤ 2.5 times ULN
  * AST or ALT ≤ 5 times ULN AND alkaline phosphatase normal
* Bilirubin normal

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No uncontrolled high blood pressure
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmia
* No New York Heart Association class III or IV heart disease

Other

* Fertile patients must use effective contraception during and for at least 3 months after study participation
* No peripheral neuropathy ≥ grade 2
* No prior severe hypersensitivity reaction to docetaxel or other drug formulated with polysorbate 80

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* No prior chemotherapy, including estramustine or suramin for prostate cancer
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 4 weeks since prior antiandrogen therapy
* No concurrent hormonal therapy except steroids for adrenal insufficiency, hormones for non-disease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* At least 8 weeks since prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* No concurrent palliative radiotherapy

Surgery

* See Disease Characteristics
* At least 4 weeks since prior surgery and recovered

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2004-06-08 (Actual); Primary Completion 2006-09-06 (Actual); Study Completion 2007-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Principal Investigator — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States